CLINICAL TRIAL: NCT06397521
Title: Gingival Margin Stability Following Esthetic Crown Lengthening by Electrocautery, Diode Laser, or a Scalpel Blade Utilizing a Double Periodontal Surgical Guide. (A Prospective Randomized Clinical Trial)
Brief Title: Gingival Margin Stability Following Esthetic Crown Lengthening Utilizing a Double Periodontal Surgical Guide
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa Adel Salah Khattab, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22879
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Crown Lengthening
Keywords: Digital; Surgical guide
MeSH Terms: interventions — Crown Lengthening

STUDY DESIGN:
Intervention Model Description: Three techniques for aesthetic crown lengthening
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scalpel crown lengthening (Experimental): Crown lengthening will be performed utilizing double periodontal surgical guide with scalpel.
  Interventions: Procedure: Crown lengthening
- Laser crown lengthening (Experimental): Crown lengthening will be performed utilizing double periodontal surgical guide with diode laser.
  Interventions: Procedure: Crown lengthening
- Electrosurgery crown lengthening (Experimental): Crown lengthening will be performed utilizing double periodontal surgical guide with electrosurgery.
  Interventions: Procedure: Crown lengthening

INTERVENTIONS:
Procedure: Crown lengthening — Investigation of the three techniques for aesthetic crown lengthening

SUMMARY:
In patients with excessive gingival display, esthetic crown lengthening procedure by means of scalpel, diode laser or electro-surgery could result in the same gingival marginal stability at 3 and 6 months follow up.

DETAILED DESCRIPTION:
Scalpel crown lengthening has been recommended as the gold standard for treating excessive gingiva. Two other established tools used for gingivectomy procedures are electrosurgery and lasers. Laser crown lengthening may have the advantages of less bleeding during the procedure, faster healing, and less pain following the procedure. Electrosurgery which involves the application of a high- frequency electric current to the gingiva has been shown to produce minimal bleeding, ease and speed of cutting and reduced postoperative pain. The null hypothesis that the three techniques for aesthetic crown lengthening (ACLP) would show equivalent gingival margin stability at 3 and 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Altered passive eruption as presence of quadratic anterior teeth [crown width/length ratio

  * 0.85 ].
* Gingival margin located coronal to the tooth cervical convexity and >2 mm of gingival band display during maximum smile.
* Patients with treated periodontal disease (i.e., stage I of periodontitis);

Exclusion Criteria:

* Patients with systemic contraindications for oral surgery as uncontrolled diabetes.
* patients on drug therapy related with drug-associated gingival enlargement.
* Areas in which the remaining amount of keratinized gingiva after the submarginal incision is less than 3 mm.
* Previous surgical treatment in the same area.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 21 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
position of the gingival margin | 3 and 6 months postoperative
  position of the gingival margin (GM) (Degree of Gingival Rebound) after performing an aesthetic crown lengthening procedure

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Adel-Khattab, PhD, Study Chair — Associate Professor Faculty of Dentistry, Ain Shams University
Locations (1):
- Doaa Adel Salah Khattab, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No